CLINICAL TRIAL: NCT01360749
Title: Multicentre, Double-Blind Trial to Evaluate the Efficacy and Safety of Lambdalina vs Placebo as an Anesthetic for Laser Hair Removal
Brief Title: Efficacy and Safety of Lambdalina (Lidocaine Cream) Versus Placebo as an Anesthetic for Laser Hair Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ISDIN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ISD-LAM-2010-01
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Local Anesthesia
Keywords: Pain management; Lidocaine
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lambdalina and placebo (Experimental): Eligible patients will receive lambdaline (lidocaine cream 40 mg/g) in Left Lower Extremity and placebo in Right Lower Extremity.
  Interventions: Drug: Lambdalina® (Lidocaine 4% cream); Drug: Placebo
- Placebo and lambdalina (Experimental): Eligible patients will receive placebo in Left Lower Extremity and lambdaline (lidocaine cream 40 mg/g) in Right Lower Extremity.
  Interventions: Drug: Lambdalina® (Lidocaine 4% cream); Drug: Placebo

INTERVENTIONS:
Drug: Lambdalina® (Lidocaine 4% cream) — Lambdaline dose: 2 g for 10 cm2.
Drug: Placebo — Placebo dose: 2 g for 10 cm2.

SUMMARY:
Double-blind, randomized, placebo-controlled trial to assess the efficacy of Lambdalina (lidocaine cream) in reducing pain associated with laser hair removal in women.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 and ≤ 65 years old.
2. Laser hair removal treatment session in the legs in the area from the knee to the ankle (first or second application).
3. Able of accomplishing the study's requirements.
4. Negative result in the pregnancy test.
5. Sterile or surgically sterilized women (hysterectomy, tubal ligation) or using adequate contraceptive methods.
6. Written informed consent prior to inclusion in the trial.

Exclusion Criteria:

- General exclusion criteria:

1. Pregnant or breastfeeding.

   - Current or previous medical conditions:
2. Skin type 5 or 6 or a history of photosensitivity.
3. Cardiovascular diseases such as unstable angina, or severe heart failure (New York Heart Association III or IV).
4. Neuropathy or paresthesia.
5. History of hepatic failure.
6. Autoimmune diseases.
7. Allergies to peanuts and/or soy and/or any components of the formulation.
8. Use or dependence on prohibited substances.
9. Other contraindications specified in the summary of product characteristics.

   - Current or previous concomitant medications:
10. Any anesthetic or analgesic treatment during 2 hours prior of study entry.
11. Concomitant treatment with antiarrhythmic drugs of class I (eg. tocainide, mexiletine) or class III (eg. amiodarone, sotalol), anticoagulants, anti-platelet aggregating and/or beta-blockers.
12. Active wounds or irritations in the area to be treated.
13. Topical treatment with corticosteroids or other topical agent in the area to be studied.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Mean change in pain intensity (Pain Visual Analogue Scale) associated to laser hair removal from baseline to the end of laser hair removal session (primary endpoint) | 30 minutes after treatment

SECONDARY OUTCOMES:
Safety assessments including AEs and SAEs | 48 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Campo Voegeli, MD, Study Chair — Clínica Dermatológica Campo De Felipe, Barcelona, Spain; Serafín Fernández, MD, Principal Investigator — Clínica Dermatológica Láser, Madrid, Spain; Antonio Campo Voegeli, MD, Principal Investigator — Clínica Dermatológica Campo De Felipe, Barcelona, Spain
Locations (2):
- Spain (2):
  - Clínica Dermatológica Campo De Felipe, Barcelona
  - Clínica Dermatológica Láser, Madrid